CLINICAL TRIAL: NCT00121784
Title: A Randomized, Open-label Study of the Effect of Replacing CNI With Sirolimus in a Standard Care Regimen of CNI, CellCept, and Steroids on Renal Function in Heart Transplant Patients
Brief Title: Heart Spare the Nephron (STN) Study - A Study of CellCept (Mycophenolate Mofetil) and Rapamune (Sirolimus) in Heart Transplant Recipients
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Poor recruitment
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MT18328
Record Dates: First submitted 2005-07-15; First posted 2005-07-21 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Heart Transplantation
MeSH Terms: interventions — Mycophenolic Acid

ARMS (1):
- 1 (Experimental): 1
  Interventions: Drug: mycophenolate mofetil [CellCept]

INTERVENTIONS:
Drug: mycophenolate mofetil [CellCept] — 1

SUMMARY:
Heart transplant patients on a standard care regimen of CNI, MMF, and corticosteroids will enter the study 4-6 weeks post-transplant. At 3 months after transplant, patients will be randomized to either continue this regimen or CNI therapy will be discontinued and replaced by sirolimus therapy (in combination with MMF and corticosteroids). The effect of these 2 regimens on efficacy, safety and renal function will be evaluated.The anticipated time on study treatment is 1-2 years and the target sample size is 500+ individuals.

ELIGIBILITY:
Inclusion Criteria:

* adult (>=18 years of age) heart transplant patients (4-6 weeks post-transplant);
* receipt of first heart (single-organ) transplant;
* standard care regimen of CNI, MMF, and corticosteroids since transplantation.

Exclusion Criteria:

* positive donor-specific cross-match at time of transplantation;
* history of malignancies, other than non-melanoma skin cancer that has been totally excised with no recurrence for 2 years;
* patients participating in another interventional clinical trial or requiring treatment with unmarketed investigational drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2005-10; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Renal function assessed by calculated GFR at 24 months post-transplant, and incidence of biopsy-proven acute rejection (BPAR) or HDC, graft loss or lost to follow-up\n

SECONDARY OUTCOMES:
Incidence of BPAR, number of episodes of BPAR per patient, time to first BPAR, incidence of re-transplant, death, rejection including antibody treated rejection, time to graft loss or death, rejection associated with HDC\n

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Chair — Hoffmann-La Roche
Locations (28):
- United States (11):
  - Chicago, Illinois
  - Maywood, Illinois
  - Boston, Massachusetts
  - Detroit, Michigan
  - Minneapolis, Minnesota
  - Cleveland, Ohio
  - Philadelphia, Pennsylvania
  - Charleston, South Carolina
  - Memphis, Tennessee
  - Dallas, Texas
  - Salt Lake City, Utah
- Australia (3):
  - Darlinghurst
  - Perth
  - Prahran
- Innsbruck, Austria
- France (7):
  - Marseille
  - Nantes
  - Paris
  - Rennes
  - Rouen
  - Tours
  - Vandœuvre-lès-Nancy
- Germany (4):
  - Berlin
  - Hanover
  - Heidelberg
  - Jena
- Spain (2):
  - Madrid
  - Pamplona